CLINICAL TRIAL: NCT05373654
Title: Observational, Prospective, Monocentric Study, Assessing the Use of Rechargeable Spinal Cord Stimulators for the Treatment of Neuropathic Pain. Quantitative and Qualitative Evaluation Protocol
Brief Title: The Use of Rechargeable Spinal Cord Stimulators for the Treatment of Neuropathic Pain
Acronym: STIMREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STIMREC; 2022-A00683-40 (Other: ANSM)
Record Dates: First submitted 2022-04-29; First posted 2022-05-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Interviews as Topic; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients that have at least one year of follow-up since the procedure. (Experimental)
  Interventions: Other: F-SUS Questionnaire; Other: Interview (only for dissatisfied patients)

INTERVENTIONS:
Other: F-SUS Questionnaire — This F-SUS questionnaire uses a Likert scale including 5 possible responses ranging from " I do not agree at all" to " I completely agree " (Celenza A 2011, Croasmun JT 2011). The F-SUS is a short questionnaire with 10 questions (Brooke J 2013). In its original version half of the questions express strong agreement and the other half disagreement. Thus, all the even-numbered items (2, 4, 6, 8, 10) allow the participant to express a very negative opinion (disagreement). On the other hand, the odd-numbered items allow the participant to express a very positive opinion (strong agreement).
Other: Interview (only for dissatisfied patients) — Patients that are dissatisfied with the recharge procedure (Score F-SUS < 70/100) will be invited to a so-called complementary information interview (an interview after the questionnaire has been completed).
  The corpus (the study group that will be interviewed) will naturally be diverse men/women, patients who were improved or not by stimulation, implanted with a rechargeable stimulator directly/replacing a stimulator, different brands of stimulator… The patient must agree to the interview and the way it will be performed (signature of consent form). The interview may be face-to -face at the site or by remote videoconference depending on the wishes and availability of the patient. There is no payment for these interviews but travelling or videoconference expenses are reimbursed All interviews will be audio- taped for further qualitative analysis.

SUMMARY:
Neuropathic pain occurs due to one or several lesions of the central or peripheral nervous system.

Spinal cord stimulation is now recommended in France by the Haute Autorité de Santé (HAS) to relieve chronic refractory neuropathic pain (HAS 2014) in the trunk, upper and lower limbs.

Spinal cord stimulation can be done either through a standard spinal cord stimulator or with a rechargeable spinal cord stimulator.

In this study, the investigators aim at assessing the recharge procedure and their constraints for consecutive patients operated for spinal cord stimulation with a rechargeable stimulator for the treatment of chronic neuropathic pain at the site by the same surgeon between 2019 and 2020.

DETAILED DESCRIPTION:
Neuropathic pain occurs due to one or several lesions of the central or peripheral nervous system. The estimated prevalence in the general population in France was 31.7% in the STOPNEP study (Study of Prevalence of Neuropathic Pain). In general, neuropathic pain becomes rapidly resistant to even specific medical treatment, and treatment by neurostimulation is increasingly common. Spinal cord stimulation is now recommended in France by the Haute Autorité de Santé (HAS) to relieve chronic refractory neuropathic pain in the trunk, upper and lower limbs.

The technique involves percutaneous or surgical placement of one or several electrodes in the epidural space to stimulate the dorsal columns of the spinal cord. The electrode is linked to a pacemaker-type stimulator which is usually placed in the subcutaneous abdominal area. Stimulation of the dorsal columns of the spinal cord is supposed to interrupt the transmission of pain messages to the areas of the brain involved in pain regulation.

The average estimated lifespan of batteries of standard stimulators is 3.7 years. This is highly dependent on the way the stimulator is used. A battery may last between 1 and 2 years in patients who use the stimulator continuously at high intensities and frequencies (above 5 volts and 60 Hz). In these cases, the stimulators must be frequently, and surgically replaced. Besides the inconvenience of repeated surgeries, the risk of infection increases with each procedure. This risk has been confirmed in patients with deep brain stimulation while the results are similar, but less clear, with spinal cord stimulation.

To prevent these problems, rechargeable stimulators have been developed and provide real medical progress for the reasons mentioned above. Rechargeable stimulators have been used in routine clinical practice since 2010. Certain rechargeable stimulators have a lifespan of 9 years, while others have a theoretically unlimited lifespan.

Thus, after more than 10 years of use of rechargeable spinal cord stimulators, the choice between a standard and rechargeable stimulator must be evaluated. The cost benefit is clear with rechargeable stimulators. However, the choice of device must also consider facility of use during daily life. The use of the rechargeable device is more complicated, mainly due to the fact that the stimulator must be recharged on a regular basis. To recharge the batteries, the patient places an antenna on the skin where the stimulator is located.

The recharge (the patient is advised to fully recharge the battery when it is at 50% capacity) can take 2 hours. When a "normal" intensity of stimulation is used (< 5 volts), the patient must charge the battery once a week, which is compatible with basically normal day to day activities. Management becomes more complicated, and even impossible in the intermediate and long term if a recharge takes longer and must be repeated more frequently, which occurs in about 25% of patients. In addition, with the most common rechargeable stimulators, the stimulator must remain constantly charged, because if it is completely empty it usually becomes impossible to recharge, requiring an intervention to replace the stimulator.

This study, observational, will consider patients for whom a rechargeable implantable spinal cord stimulator was placed as part of standard of care, at least one year ago.

The main goal is to determine the proportion of patients who are dissatisfied with the recharge procedure after at least one year of use, and to evaluate their experience to determine the causes of their dissatisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women implanted with a rechargeable spinal cord stimulator in 2019 and 2020,
2. Implantation carried out more than one year before the date of inclusion in the study,
3. Primary implantation of a rechargeable spinal cord stimulator or replacement of a non-rechargeable spinal cord stimulator with a rechargeable spinal cord stimulator,
4. Dorsal or cervical spinal cord stimulation,
5. Patient operated by the same surgeon,
6. Patient informed of the study and consented to take part.

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Patient whose cognitive abilities, as assessed by the investigator, do not allow them to complete the F-SUS questionnaire or the numerical pain scale.
3. Patient covered by legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients dissatisfied with the recharge procedure after at least one year of use. | Up to 1 year
  F-SUS Questionnaire. This questionnaire uses a Likert scale including 5 possible responses ranging from " I do not agree at all" to " I completely agree ". The F-SUS is a short questionnaire with 10 questions. The total maximum score is 100. The total score will be used for the different analyses because the F-SUS is considered to be a unidimensional score. Satisfaction will be considered to be good with a score of 70 and excellent with 90. Satisfaction is correct between 50 and 70 (indicating that the system needs to be improved). At a score below 50 the system is unusable.
Evaluation of dissatisfied patients' experience to determine the causes of their dissatisfaction. | Up to 1 year
  Interview

SECONDARY OUTCOMES:
Comparison of numerical pain scale before spinal cord stimulator surgery and at least one year after the surgery. | Up to 1 year
  The analgesic result of the spinal cord stimulation will be evaluated with a numerical pain scale ranging from 0 ("No pain") to 10 ("Maximum imaginable pain"). The value that will be compared to the preoperative numerical pain scale will be the mean of 3 measurements obtained on the day (morning, noon, night) before the questionnaire is filled out.
Comparison of patients' satisfaction between different stimulators models. | Up to 1 year
  The brand of rechargeable stimulator will be collected for the study. The satisfaction level will be established with the F-SUS questionnaire. This questionnaire uses a Likert scale including 5 possible responses ranging from " I do not agree at all" to " I completely agree ". The F-SUS is a short questionnaire with 10 questions. The total maximum score is 100. The total score will be used for the different analyses because the F-SUS is considered to be a unidimensional score. Satisfaction will be considered to be good with a score of 70 and excellent with 90. Satisfaction is correct between 50 and 70 (indicating that the system needs to be improved). At a score below 50 the system is unusable.
Patients' satisfaction | During the year following qualitative analysis.
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Brétéché, Nantes, France

REFERENCES:
- [Background] Moisset X, Bouhassira D, Attal N. French guidelines for neuropathic pain: An update and commentary. Rev Neurol (Paris). 2021 Sep;177(7):834-837. doi: 10.1016/j.neurol.2021.07.004. Epub 2021 Jul 28. PMID 34332778
- [Background] Bouhassira D, Lanteri-Minet M, Attal N, Laurent B, Touboul C. Prevalence of chronic pain with neuropathic characteristics in the general population. Pain. 2008 Jun;136(3):380-387. doi: 10.1016/j.pain.2007.08.013. Epub 2007 Sep 20. PMID 17888574
- [Background] Cameron T. Safety and efficacy of spinal cord stimulation for the treatment of chronic pain: a 20-year literature review. J Neurosurg. 2004 Mar;100(3 Suppl Spine):254-67. doi: 10.3171/spi.2004.100.3.0254. PMID 15029914
- [Background] Dones I, Levi V. Spinal Cord Stimulation for Neuropathic Pain: Current Trends and Future Applications. Brain Sci. 2018 Jul 24;8(8):138. doi: 10.3390/brainsci8080138. PMID 30042314
- [Background] Blackburn AZ, Chang HH, DiSilvestro K, Veeramani A, McDonald C, Zhang AS, Daniels A. Spinal Cord Stimulation via Percutaneous and Open Implantation: Systematic Review and Meta-Analysis Examining Complication Rates. World Neurosurg. 2021 Oct;154:132-143.e1. doi: 10.1016/j.wneu.2021.07.077. Epub 2021 Jul 31. PMID 34343680
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Meyerson BA, Linderoth B. Mode of action of spinal cord stimulation in neuropathic pain. J Pain Symptom Manage. 2006 Apr;31(4 Suppl):S6-12. doi: 10.1016/j.jpainsymman.2005.12.009. PMID 16647596
- [Background] Echeverria-Villalobos M, Mitchell J, Fiorda-Diaz J, Weaver T. Effects of Dorsal Column Spinal Cord Stimulation on Neuroinflammation: Revisiting Molecular Mechanisms and Clinical Outcomes on Chronic Lumbar/Leg Pain and Failed Back Surgery Syndrome. J Pain Res. 2021 Jul 30;14:2337-2345. doi: 10.2147/JPR.S309872. eCollection 2021. PMID 34354373
- [Background] Lam CK, Rosenow JM. Patient perspectives on the efficacy and ergonomics of rechargeable spinal cord stimulators. Neuromodulation. 2010 Jul;13(3):218-23. doi: 10.1111/j.1525-1403.2009.00269.x. Epub 2010 Feb 24. PMID 21992835
- [Result] Costandi S, Mekhail N, Azer G, Mehanny DS, Hanna D, Salma Y, Bolash R, Saweris Y. Longevity and Utilization Cost of Rechargeable and Non-Rechargeable Spinal Cord Stimulation Implants: A Comparative Study. Pain Pract. 2020 Nov;20(8):937-945. doi: 10.1111/papr.12926. Epub 2020 Jul 27. PMID 32543118
- [Result] Pepper J, Zrinzo L, Mirza B, Foltynie T, Limousin P, Hariz M. The risk of hardware infection in deep brain stimulation surgery is greater at impulse generator replacement than at the primary procedure. Stereotact Funct Neurosurg. 2013;91(1):56-65. doi: 10.1159/000343202. Epub 2012 Nov 29. PMID 23207787
- [Result] Hoelzer BC, Bendel MA, Deer TR, Eldrige JS, Walega DR, Wang Z, Costandi S, Azer G, Qu W, Falowski SM, Neuman SA, Moeschler SM, Wassef C, Kim C, Niazi T, Saifullah T, Yee B, Kim C, Oryhan CL, Rosenow JM, Warren DT, Lerman I, Mora R, Hayek SM, Hanes M, Simopoulos T, Sharma S, Gilligan C, Grace W, Ade T, Mekhail NA, Hunter JP, Choi D, Choi DY. Spinal Cord Stimulator Implant Infection Rates and Risk Factors: A Multicenter Retrospective Study. Neuromodulation. 2017 Aug;20(6):558-562. doi: 10.1111/ner.12609. Epub 2017 May 11. PMID 28493599
- [Result] Falowski SM, Provenzano DA, Xia Y, Doth AH. Spinal Cord Stimulation Infection Rate and Risk Factors: Results From a United States Payer Database. Neuromodulation. 2019 Feb;22(2):179-189. doi: 10.1111/ner.12843. Epub 2018 Aug 17. PMID 30117635
- [Result] Van Buyten JP, Fowo S, Spincemaille GH, Tronnier V, Beute G, Pallares JJ, Naous H, Zucco F, Krauss JK, De Andres J, Buchser E, Costantini A, Lazorthes Y. The restore rechargeable, implantable neurostimulator: handling and clinical results of a multicenter study. Clin J Pain. 2008 May;24(4):325-34. doi: 10.1097/AJP.0b013e31816216a9. PMID 18427231